CLINICAL TRIAL: NCT06046170
Title: Adaptation and Feasibility of the Community-Based Anxiety Program Tailored for Autism (CAPTA): A Randomized Control
Brief Title: Adaptation and Feasibility of the Community-Based Anxiety Program Tailored for Autism (CAPTA)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Pennsylvania (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Eric A Storch, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-54327
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Autism Spectrum Disorder; Separation Anxiety; Generalized Anxiety Disorder; Social Anxiety Disorder of Childhood
Keywords: cognitive behavioral therapy; children; adolescents; anxiety; Community mental health clinics
MeSH Terms: conditions — Anxiety Disorders; Autism Spectrum Disorder; Anxiety, Separation; Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized assignment to one of two conditions
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Active Comparator): Participants will receive cognitive behavioral therapy that has been adapted for autistic youth with anxiety. These sessions will also include components of exposure. Participants will receive therapy around once a week for 14 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Treatment as Usual (Placebo Comparator): Participants will complete treatment as usual. They will be referred to other community resources, including skills training. Additionally, participants may begin or end therapy and/or medication.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants will receive cognitive behavioral therapy with elements of exposure in order to target anxious behaviors.
  Arms: Cognitive Behavioral Therapy
Other: Treatment as Usual — Participants will receive treatment as usual at a community mental health center, including receiving skills training.
  Arms: Treatment as Usual

SUMMARY:
Anxiety is very common in autistic youth. Recently, an intervention has been created by the investigators to target these symptoms in autistic youth in a community setting. The purpose of this study is to determine the feasibility of implementing this treatment in community care centers.

DETAILED DESCRIPTION:
As many as 50% of autistic youth have at least 1 anxiety disorder. Cognitive-behavioral therapy (CBT) for autistic youth is effective at treating anxiety, but access is limited. The investigators have tailored the treatment to make it more accessible to families in the participants' home communities. The purpose of this project is to investigate how feasible it is to implement Community-Based Anxiety Programs Tailored for Autism (CAPTA) in community settings.

ELIGIBILITY:
Inclusion Criteria:

1. The adolescent is between the ages of 7 to 17 upon enrollment with an established autism spectrum disorder diagnosis (ASD) made by a standardized assessment (e.g., Autism Diagnostic Observation Schedule-Second Edition; Childhood Autism Rating Scale-Second Edition), confirmed by the Social Communication Questionnaire (SCQ) ≥ 11 and/or total score ≥ 7 on the Autism Diagnostic Observation Schedule-2 (ADOS-2). Dr. Storch will review diagnostic reports to determine whether an appropriate ASD diagnosis has been established.
2. The adolescent has clinically elevated symptoms of anxiety based on elevated scores on the Pediatric Anxiety Rating Scale modified for Autism Spectrum Disorder (>12).
3. Anxiety is the primary concern and the child is appropriate for intervention focus, as determined by completion of a structured psychiatric diagnostic interview (the Mini International Neuropsychiatric Interview) by an independent evaluator (IE) supervised by an experienced, licensed psychologist determines that the child is appropriate for the intervention focus.
4. Child has a verbal intelligence quotient greater than or equal to 70, as measured by the Verbal Comprehension Index of the Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V).
5. One parent/guardian is able and willing to participate (i.e., available during therapy sessions, attend study assessments).
6. Child is eligible to receive services at the participating clinic.
7. Both parent and child can read and/or understand English and/or Spanish.
8. Both parent and child reside in Texas or Pennsylvania.

Exclusion Criteria:

* 1.) The child has a diagnosis of psychotic disorder as determined by completion of a structured psychiatric diagnostic interview (the Mini International Neuropsychiatric Interview).

  2.) The child has severe current suicidal/homicidal ideation and/or self-injury requiring medical intervention (referrals will be made for appropriate clinical intervention).

  3.) The child is receiving concurrent psychotherapy for anxiety.

  4.) If child is taking psychotropic medication, regimen must have been started 8 weeks ago and stable for the past 4 weeks (or 2 weeks for stimulants or benzodiazepines). If appropriate, a delayed entry will be allowed so that once a child is on a stable dosage s/he may be enrolled.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale - ASD | baseline (before treatment), during treatment (on average 14 weeks), post-treatment (last week of treatment), 3 month follow up
  Clinician-rated child anxiety severity throughout the past week. Each item is scored on a 0 to 5 scale (higher scores correspond to greater severity), yielding a total between 0 and 35. This measure has been modified for autistic youth

SECONDARY OUTCOMES:
Anxiety Disorders Interview Schedule (ADIS-IV) with Clinical Severity Ratings | baseline (before treatment), during treatment (on average 14 weeks), post-treatment (last week of treatment), 3 month follow up
  Clinician-rated diagnostic interview that includes current anxiety disorders, depression, obsessive-compulsive disorder, and related disorders. Each diagnostic category is coded as present or absent based on symptom criteria and clinical severity ratings (CSRs), which indicate the level of clinical interference. CSRs are scored on a 0-8 scale (0 = not at all; 8 = very, very much). CSRs of 4 or above indicate the clinical levels.
Clinical Global Impression-Improvement | baseline (before treatment), during treatment (on average 14 weeks), post-treatment (last week of treatment), 3 month follow up
  Clinician-rated child psychopathology severity rating. A single item is scored 0-6 (0= very much improved; 6= very much worse).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No